CLINICAL TRIAL: NCT07402733
Title: PIC Rehab: Psychologically Informed Cervicovestibular Rehabilitation for Mild Traumatic Brain Injury: A Feasibility Trial
Brief Title: Psychologically Informed Cervicovestibular Rehabilitation (PIC Rehab) for Mild Traumatic Brain Injury: A Feasibility Trial
Acronym: PIC Rehab
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sport Injury Prevention Research Centre (Other)
Collaborators: University of Calgary (Other); Brain Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIC Rehab
Record Dates: First submitted 2026-01-28; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mild Traumatic Brain Injury, Concussion
Keywords: rehabilitation; cervical spine; vestibular; cognitive behavioural therapy; treatment
MeSH Terms: conditions — Brain Concussion | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: This study is a pilot feasibility study where the initial group will receive standard cervicovestibular rehabilitation. Subsequently, the same therapists will be trained in psychologically informed cervicovestibular rehabilitation and the patients recruited after this training will be in the psychologically informed cervicovestibular rehabilitation group.
Who Masked: Participant
Masking Description: Participants will be blinded to the hypothesis of the study and to the opposite treatment group to which they are assigned. Thus, two separate consent forms will be used in the study - one for each type of treatment received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervicovestibular Rehabilitation (CVPT) (Active Comparator): CVPT includes treatments targeting neuromuscular and sensorimotor control in combination with manual therapy and soft tissue techniques as indicated.5 16 Specific rehabilitation exercises are gradually progressed, performed in combination with symptom-tolerated aerobic exercise, and eventually evolve to task, context, and/or sport specific exercises.16 From a mechanistic standpoint, the goal of this treatment is to facilitate sensorimotor integration (i.e. integration of visual, vestibular, proprioceptive input and resultant motor output) and either reweigh central balancing of stimuli to optimize function of these systems or upregulate the use of alternate systems in the event that one of the sensory systems is not optimally operating.5 17 Recent international consensus recommendations and clinical practice guidelines recommend CVPT as a treatment that has some of the strongest evidence to date to facilitate recovery.14 18
  Interventions: Behavioral: Cervicovestibular Rehabilitation (CVPT)
- Psychologically Informed CVPT (PIC Rehab) (Experimental): Cognitive behavioural therapy (CBT) is a form of treatment that uses multiple non-pharmacological strategies including education, behavioural and cognitive strategies to assist with decreasing symptoms. The experimental PIC Rehab arm will include principles of CBT in combination with the CVPT.
  Interventions: Behavioral: Psychologically Informed CVPT (PIC) Rehab; Behavioral: Cervicovestibular Rehabilitation (CVPT)

INTERVENTIONS:
Behavioral: Psychologically Informed CVPT (PIC) Rehab — Arm Description: Cognitive behavioural therapy (CBT) is a form of treatment that uses multiple non-pharmacological strategies including education, behavioural and cognitive strategies to assist with decreasing symptoms. The experimental PIC Rehab arm will include principles of CBT in combination with the CVPT.
  Arms: Psychologically Informed CVPT (PIC Rehab)
Behavioral: Cervicovestibular Rehabilitation (CVPT) — Cervical and vestibular rehabilitation including individually targeted impairments based treatment techniques such as neuromuscular control, joint position sense, manual therapy, adaptation, habituation, canalith repositioning maneouvers, standing balance exercises, dynamic balance exercises, sport and work specific exercises.

SUMMARY:
Mild traumatic brain injuries ("mTBIs") affect over 480,000 Canadians each year. While many individuals recover in the initial 4 weeks following mTBI, in up to 30% of individuals symptoms and functional impairments often persist leading to significant disability, decreased quality of life and participation in education, physical and occupational related activities. An assessment that evaluates multiple systems is recommended for individuals with mTBI, often involving multiple health care professionals to assess different areas of function (e.g. oculomotor, vestibular, balance, mood, cognition, etc). Current evidence supports the use of cervicovestibular rehabilitation (CVPT) (which includes physiotherapy techniques aimed at treating the neck, balance, visual and other sensory systems) and symptom-tolerated exercise. Evidence suggests that collaborative care, cognitive behavioural therapy (CBT) may be of benefit. However, the added value of CVPT and CBT in combination co-designed by patients and community partners has not yet been evaluated in mTBI. In other pain and dizziness conditions, the addition of CBT to physical/vestibular rehabilitation yielded improved outcomes. Here we take a transdisciplinary team-based approach to evaluate an integrated combination of CVPT and CBT.

This study will recruit a total of 34 people ages 18-70 years old who have ongoing symptoms following an mTBI for more than two weeks. The first 17 patients will receive CVPT along and the second 17 patients will receive psychologically informed CVPT ("PIC" Rehab). This study will help determine if combined therapy has an additive effect on helping patients recovery from mTBI.

DETAILED DESCRIPTION:
Problem: Mild traumatic brain injuries and concussions affect over 480,000 or 1.2% of Canadians each year.1-3 While many individuals recover in the initial 4 weeks following mTBI, up to 30% have persisting symptoms and functional impairments, leading to significant disability, decreased quality of life, and reduced participation in education, physical, and occupational related activities.

Dizziness, balance problems, headaches, and neck pain: Headaches and dizziness are consistently the most commonly reported symptoms following mTBI with estimates of up to 95% of individuals reporting headaches and 40-80% reporting dizziness. In a majority of cases, these symptoms are reported concurrently. Standing balance and dynamic balance deficits have consistently been identified following mTBI, some of which resolve early post-injury (within 3-5 days), while some balance problems remain for weeks to months following injury. Dizziness, balance problems, headaches, and neck pain are associated with greater odds of developing persisting symptoms. In addition, persisting dizziness, headaches, neck pain, and balance impairments can lead to decreased participation in recreational, social, occupational, and educational activities as well as lower quality of life. Decreased activity can, in turn, lead to significant morbidity due to secondary health complications. Therefore, treatments aimed at minimizing headaches, dizziness and balance problems following mTBI are urgently needed to minimize the public health burden of this commonly occurring injury.

Treatment of dizziness, balance problems, headaches, and neck pain following mTBI: Previous randomized controlled trials (RCTs) have identified large positive treatment effects following targeted cervical and vestibular rehabilitation (CVPT) for children, adolescents, and adults with dizziness, neck pain, and headaches following mTBI. These treatments are personalized, based on the individual's profile of specific impairments. CVPT includes treatments targeting neuromuscular and sensorimotor control in combination with manual therapy and soft tissue techniques as indicated. Specific rehabilitation exercises are gradually progressed, performed in combination with symptom-tolerated aerobic exercise, and eventually evolve to task, context, and/or sport specific exercises. From a mechanistic standpoint, the goal of this treatment is to facilitate sensorimotor integration (i.e. integration of visual, vestibular, proprioceptive input and resultant motor output) and either reweigh central balancing of stimuli to optimize function of these systems or up-regulate the use of alternate systems in the event that one of the sensory systems is not optimally operating. Recent international consensus recommendations and clinical practice guidelines recommend CVPT as a treatment that has some of the strongest evidence to date to facilitate recovery. However, up to 27% of individuals may not respond to CVPT5, necessitating other treatment options.

Cognitive Behavioural Therapy: For individuals with persisting symptoms following mTBI, evidence supports the use of cognitive behavioural therapy (CBT). CBT is a form of treatment that uses multiple non-pharmacological strategies including education, behavioural and cognitive strategies. This form of non-pharmacological treatment has demonstrated safety and efficacy for a number of different conditions including insomnia, depression, mental health, and more recently for mTBI. For individuals with chronic pain, improvements in anxiety and depressive symptoms have been demonstrated but no difference in pain intensity or pain catastrophizing has been found to date. Patient centred approaches are necessary to optimize effectiveness. In individuals with dizziness, the addition of CBT to physical and/or vestibular rehabilitation may yielded improved outcomes.

Thus, CVPT and CBT in combination may have additive effects for individuals with mTBI. Here we take a transdisciplinary team-based approach to evaluate an integrated combination of CVPT and CBT.

Objectives:

We will conduct a pilot trial using a stepped approach to evaluate the feasibility and patient perceptions of CVPT alone as compared to CVPT in combination with CBT (hereafter referred to as PIC Rehab, or psychologically-informed CVPT) on 1) symptom severity and 2) time to resolution of mTBI related symptoms in adults with symptoms for greater than 14 days following mTBI.

The specific objectives of this study are as follows:

Objective 1: Determine the feasibility of PIC Rehab; Objective 2: Generate preliminary estimates of effect for PIC Rehab on mTBI related symptom resolution compared to CVPT alone; Objective 3: Describe changes by sex in domain specific outcomes of PIC Rehab compared to CVPT alone.

We hypothesize that PIC Rehab will be feasible and will have a greater impact on resolution of symptoms for participants with concomitant anxiety, depression, patient specific functional disability, than CVPT alone.

Methods:

Thirty-four adults aged 18-70 years with symptoms of dizziness, neck pain and/or headaches for at least 14 days following mTBI who are referred for cervicovestibular physiotherapy with one or more impairments related to the vestibular, oculomotor, sensorimotor, cervical spine, neuromuscular control, will be invited to participate. The participants who are included in this study are those with impairments that have previously been shown to respond to cervicovestibular rehabilitation. Patients who have previously undergone a session of cervicovestibular physiotherapy will be excluded from the study. The first 15 participants will complete typical CVPT and the next "step" of the study will have the following 15 participants complete PIC Rehab. Participants will be recruited consecutively in the order they are referred/approached based on their initial symptom reports of headaches, dizziness and/or neck pain at the time of presentation to the clinic, inclusive of both sexes and all genders, with the aim to have equal numbers of male and female participants.

Participants will be eligible for participation if they are referred to or seek treatment at Evidence Sport and Spinal Therapy for cervicovestibular rehabilitation following mTBI. For the purposes of this pilot feasibility trial we will limit our recruitment to one clinic with multiple therapists to enable future study of a larger trial at multiple clinics and, thus, avoid the chance of contamination between control and intervention groups. Consent to contact will be obtained in clinic for those patients meeting the inclusion criteria as part of the initial intake to the clinic and a member of the research team will follow-up and contact the patient by phone.

Eligibility Screen: Patients who agree to be contacted will undergo an eligibility screen with questionnaires (e.g., PCSS) by telephone with a research assistant. If the patient meets the eligibility for the trial they will then be sent a consent form to review and sign online followed by the initial demographic forms, questionnaires and subsequently scheduled for the initial assessment. After completing the initial assessment, the RA will confirm eligibility. It is possible that participants may have pre-existing relationships with the researchers or clinicians that are part of the research team as participants will be recruited through community sport medicine and/or physiotherapy clinics. Thus, all potential participants will be made aware that their choice to participate in this study will in no way affect the care that they receive and that they are free to decline participation at any time.

Protocol:

Participants will be blinded to the hypothesis of the study and to the opposite treatment group to which they are assigned. Thus, two separate consent forms will be used in the study - one for each type of treatment received. Both treatment groups will be seen once weekly for 8 weeks or until the time of symptom resolution and medical clearance to return to sport/learn/occupation and outcomes will be repeated at the 8 week time point. All of the physiotherapists who are participating in the study will undergo a standard CVPT training course. Following recruitment of the initial 15 patients, all therapists will undergo and online and in person training course for PIC Rehab. To facilitate recruitment in a timely fashion and prevent delays between arms, the first 3 of 6 therapists who complete treatment with their participants will complete the PIC Rehab training and the second 3/6 will complete a later training course for PIC Rehab.

CVPT alone: The control intervention will be the typical standard of care of CVPT (Schneider et al 2014, 2018) including individualized cervical and vestibular rehabilitation based on the patient's presentation, including symptom-tolerated exercise.

PIC Rehab: The Psychological Informed-CVPT (PIC Rehab) intervention (modified from Herdman et al) will include education, goal setting, distraction techniques, reattribution of symptoms, relaxation, in vivo exposure, cognitive therapy and problem solving. Collaborative training for physiotherapist providing the PIC Rehab will occur with the study team (KS, NS, KOY, CP).

The stepped process of the treatments will minimize contamination by therapist knowing the principles of the PIC Rehab. Adherence to the intervention will be assessed using scheduled audio recordings of the treatment sessions (to measure therapist adherence to the protocol) and patient reports of completion of home exercises (patient adherence). As this is a pilot feasibility study, a sample of 30 participants (15 in each group) allowing for two drop outs per group based on previous studies done at our centre was deemed to be pragmatic with in a 6 month time frame.

Initial Assessment: The initial assessment will take approximately 90 minutes and participants will complete a series of in person outcomes with the study physiotherapist as listed below that are specific to domains that may be affected by concussion. Where relevant, additional questions and health history information and clinically relevant outcomes will be gathered in keeping with the current standard of care.

Follow-up appointments: All participants will complete a brief set of questionnaires on REDCap at the time of each follow-up appointment to capture current symptoms, completion of home program exercises and any additional treatment that has been undertaken since the time of the previous appointment. In the event that new symptoms are present, the relevant self report and in person clinical outcomes related to the specific symptoms will be repeated. Treating physiotherapists will complete an adherence questionnaire after each session and record all subcomponents of treatment individualized to the patient.

Outcome assessments: Outcome assessments, both self report and in person clinical outcomes, will be repeated 8 weeks after the initial baseline assessment. Following participation in the trial, participants and therapists will be invited to take part in semi-structured interviews to share their experiences as part of the trial, including barriers and facilitators to the rehabilitation protocols.

Outcomes:

Primary feasibility outcomes will include recruitment, retention rate, adverse events, clinical implementation barriers and facilitators faced, and adherence to protocol (therapist).

Secondary outcomes of recovery including time to resolution of symptoms (days) to inform a phase 2 clinical trial. In keeping with international recommendations, and exploratory outcomes that assess impairment specific factors that may change with treatment (i.e. cervical spine, vestibulo-ocular, dynamic balance, etc) will be included.

Secondary outcomes will include change in symptom severity scores on the PCSS (/132), time to resolution of symptoms (days), time to medical clearance to return to sport, learn and work (days) (as relevant) to inform a phase 2 clinical trial. These outcomes will be defined as per the latest international consensus recommendations (page 702). Return to work (RTW) will be defined in the same was as return-to-learn and will be defined as: return to pre-injury occupational activities with no new support, including occupational accommodations or modifications.

Exploratory outcomes are outcomes that are part of typical clinical care and will include impairment based/domain specific outcomes that are the current best available outcomes and aligned with previous trials in the area. All outcomes will also be described by sex. Exploratory outcomes will include the following:

* Fear Avoidance Behaviour after Traumatic Brain Injury Questionnaire (FAB-TBI)
* World Health Organization Disability Assessment Schedule (WHODAS) 2.0 12 item self-report version
* Anxiety (Generalized Anxiety Disorder-7, GAD-7)
* Depression (Personal Health Questionnaire-9, PHQ-9)
* Sleep Screen
* Post Concussion Symptom Scale from the Sport Concussion Assessment Tool 6 (SCAT6)
* Test of Memory Malingering (TOMM)
* Dizziness Handicap Inventory
* Modified Dizziness Questionnaire
* Neck Disability Index
* Neck Pain Questionnaire
* Patient Specific Functional Scale (PSFS)
* Post Traumatic Headache Questionnaire
* Subjective Units of Discomfort Scale (SUDS)
* Neurological screen including cranial nerve, cerebellar and long track signs
* Cervical Spine: Cervical Spine range of motion, cervical flexor endurance, cervical flexion rotation test, craniocervical flexion test, manual spinal examination, palpation for segmental tenderness, extension rotation test, palpation of tender trigger points, palpation of greater and lesser occipital nerves
* Tests done with fixation removed including spontaneous nystagmus, gaze evoked, fixation, hyperventilation, intracranial pressure, head shaking, positional testing (including Dix-Hallpike and Roll tests right and left).
* Vestibulo-ocular reflex tests: head thrust test, dynamic visual acuity
* Quantified Vestibular Ocular Motor Screen (qVOMS)
* Motion sensitivity Test
* Dynamic Balance: functional gait assessment (FGA) and advanced FGA
* Balance Error Scoring System (BESS)
* Buffalo Concussion Treadmill Test (BCTT) or Bike Test (BCBT) as appropriate depending on the patient preference
* Orthostatic Vital Signs

Data Analysis:

Primary feasibility outcomes will be summarized using descriptive statistics [means (standard deviations) or medians/modes (ranges or interquartile ranges) or proportions] as appropriate. Secondary outcomes will be summarized descriptively by treatment group. In addition, exploratory Kaplan Meier survival analysis curves will be constructed by group for time to resolution of symptoms, return to sport, learn, occupation will be evaluated using Kaplan Meier survival analysis curves with the outcome of 8 weeks. Exploratory outcomes will be described by treatment group and sex using descriptive statistics as appropriate based on the outcome and the distribution of the data. Thematic analysis will be used to evaluate barriers and facilitators to PIC Rehab for both participants and providers.

ELIGIBILITY:
Inclusion Criteria:

* Reporting dizziness, neck pain and/or headaches for at least 14 days following mild traumatic brain injury/concussion who are referred for cervicovestibular physiotherapy with one or more impairments related to the vestibular, oculomotor, sensorimotor, cervical spine, neuromuscular control.

Exclusion Criteria:

* Patients who have previously undergone a session of cervicovestibular physiotherapy will be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment | From enrollment to the end of treatment at 8 weeks.
  Number of participants recruited
Feasibility - retention rate | From enrolment to the end of treatment at 8 weeks
  Number of participants completing the trial divided by the total number of participants recruited
Feasibility - Adverse events | From enrolment to the end of treatment at 8 weeks
  Total number of adverse events
Feasibility - barriers and facilitators | From enrolment to the end of treatment at 8 weeks.
  Barriers and facilitators to the protocol as described by the participants and the physiotherapists.
Feasibility - Adherence to protocol by therapist | From enrolment to the end of treatment at 8 weeks.
  Adherence will be measured through voice recording review of the therapist treatment prescription in comparison to the specific group treatment protocol. The choice of treatment by the therapist will be matched to the treatment choice on the treatment protocol and rated as "yes" adheres or "no" does not adhere for each component of treatment at each recorded session. The proportion of components adhered to will be summarized.

SECONDARY OUTCOMES:
Symptom Severity Score (SSS) | Initial and 8 weeks
  As measured on the Post Concussion Symptom Scale from the Sport Concussion Assessment tool, /132 where 0 represents no symptoms and 132 the most severe symptoms
Date of Medical Clearance to Return to Sport | From enrolment until treatment completion at 8 weeks
  Defined as per the Amsterdam International Consensus statement (Patricios, Schneider et al 2023, page 702): "Completion of the RTS strategy with no symptoms and no clinical findings associated with the current concussion at rest and with maximal physical exertion."
Date of Return to full learn | From enrolment to the end of treatment at 8 weeks.
  Defined as per the Amsterdam international consensus on concussion in sport (Patricios, Schneider et al 2023 page 702): Return to pre-injury learning activities with no new academic support, including school accommodations or learning adjustments.
Return to work | From enrolment to end of treatment at 8 weeks
  Return to pre-injury occupational activities with no new support, including occupational accommodations or modifications

OTHER OUTCOMES:
Exploratory - Fear Avoidance Behaviour after Traumatic Brain Injury Questionnaire (FAB-TBI) | Initial and 8 weeks
  Validated measures of fear avoidance in TBI, 0-48 with higher score representing greater fear avoidance.
Exploratory - World Health Organization Disability Assessment Schedule (WHODAS) 2.0 12 item | Initial and 8 weeks following treatment initiation
  WHO measure of self reported disability, scored 0-48 with higher score representing greater disability.
Exploratory - Generalized Anxiety Disorder - 7 | Initial and 8 weeks following treatment initiation
  GAD-7 to measure self reported anxiety, scored 0-21 with greater score representing anxiety
Exploratory - Personal Health Questionnaire-9 | Initial and 8 weeks following treatment initiation
  Personal Health Questionnaire - 9 to screen for depression, 0-27 with higher scores representing greater depression severity
Exploratory - Test of Memory Malingering (TOMM) | Initial to 8 weeks following treatment initiation
  Validated test to evaluate for malingering, scores of 0-50 with scores less than 45 indicative of insufficient effort.
Exploratory - Dizziness Handicap Inventory (DHI) | Initial to 8 weeks following treatment initiation
  25 item self report outcome measure to evaluate self perceived dizziness disability, scores range of 0-100 with greater scores indicative of greater perceived disability due to dizziness.
Exploratory - Modified Dizziness Questionnaire | Initial to 8 weeks following treatment initiation
  Self reported characteristics of dizziness outcome including nature, duration, aggravating and easing factors with items checked as "yes" used to categorize dizziness.
Exploratory - Neck Disability Index (NDI) | Initial to 8 weeks following treatment initiation
  Self reported outcome to describe characteristics of neck disability, scored 0-50 with greater scores indicating greater neck disability
Exploratory - Patient Specific Functional Scale (PSFS) | Initial to 8 weeks following treatment initiation
  Self reported difficulty scale for 3-5 specific functional activities that affect the individual patient. Each individual item is rated 0-10 with greater scores indicate more difficulty with function on the specific activity and 0 representing no difficulty.
Neurological Screen findings | Initial and 8 weeks following treatment initiation
  Any findings of cranial nerve, cerebellar or other long track signs, rated as present/absent
Cervical spine range of motion | Initial and 8 weeks following treatment initiation
  Cervical spine range of motion full/reduced
Cervical flexor endurance | Initial and 8 weeks following treatment initiation
  Time (seconds) the participant is able to lift and hold there head per Schneider et al 2018
Cervical flexion rotation test | Initial and 8 weeks following treatment initiation
  Test to evaluate upper cervical spine involvement, positive/negative
Craniocervical flexion test | Initial and 8 weeks following treatment initiation
  Evaluates craniocervical flexion ability, mmHg with a range of 20-30mmHg and greater scores indicating better performance.
Manual spinal exam | Initial and 8 weeks following treatment initiation
  Evaluation of segmental pain rated as positive if >3/10 pain is reproduced and limited motion
Palpation for segmental tenderness | Initial and 8 weeks following treatment initiation
  rated as positive if reproduced familiar pain with palpation of deep structures segmentally >3/10
Extension rotation test | Initial and 8 weeks following treatment initiation
  Rated as positive if reproduction of familiar pain >3/10 with extension and rotation of cervical spine
Palpation of tender trigger points | Initial and 8 weeks following treatment initiation
  Reproduction of pain with palpation of tender trigger points yes/no
Greater and lesser occipital nerve findings | Initial and 8 weeks following treatment initiation
  Palpation of greater and/or lesser occipital nerve reproducing familiar pain, yes/no
Dix-Hallpike test | Initial and 8 weeks following treatment initiation
  Positional test positive for BPPV posterior or anterior canal; rated as positive/negative
Nystagmus identified with fixation removed | Initial and 8 weeks following treatment initiation
  Tests done with videonystagmography identify nystagmus, categorized according to test findings; rated as present/absent and if present, further categorized by direction (e.g. right beat, up beat)
Head thrust test | Initial and 8 weeks following treatment initiation
  Also called head impulse test, positive/negative to suggest potential altered vestibulo-ocular reflex function
Dynamic visual acuity | Initial and 8 weeks following treatment initiation
  Evaluates the difference between head still and head moving using an Early Test for Diabetic Retinopathy (ETDRS) chart, logMAR with greater change indicating worse performance with head motion
Vestibular Ocular Motor Screen (VOMS) | Initial and 8 weeks following treatment initiation
  As per Mucha et all, symptom reproduction of >2/10 with at least two of the included 7 vestibular and oculomotor tests and/or near point of convergence >6cm.
Functional gait assessment | Initial and 8 weeks following treatment initiation
  Evaluates dynamic balance in a series of 10 different tests, /30 with greater scores indicating better balance performance, range 0-30
Balance Error Scoring System | Initial and 8 weeks following treatment initiation
  Measure of standing balance on floor and on foam (where safe and appropriate) in three conditions: Romberg, tandem, single leg stance. /30 for each of foam and floor, with better balance with less errors reported (i.e. lower score), range 0-30
Maximum heart rate attained on Buffalo Concussion Treadmill Test or Bike Test | Initial and 8 weeks following treatment initiation
  measure of physical exertion, mode of test determined by patient preference
Presence of orthostatic intolerance | Initial and 8 weeks following treatment initiation
  symptom reproduction with change from supine to stand with at least one of drop in systolic BP of >=20mmHg, diastolic >=10mmHg, HR decrease or HR increases >=30bpm (per Patricios et al 2023)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schneider, PT PhD, Principal Investigator — University of Calgary
Locations (1):
- Evidence Sport and Spinal Therapy North, Calgary, Alberta, Canada